CLINICAL TRIAL: NCT00595608
Title: Sterimar vs Saline Sprays in Nasal Surgical Aftercare - a Blinded, Randomised Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: NHS Grampian, R&D department, NHS Grampian
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07/S0802/45; 07/S0802/45
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2007-12

CONDITIONS: Nasal Surgery
Keywords: aftercare; nasal septum; turbinates
MeSH Terms: interventions — Salts; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Nasal Sterimar spray
  Interventions: Drug: Sterimar Spray
- 2 (Active Comparator): Nasal saline spray
  Interventions: Drug: Generic homemade nasal saline spray (salt and water)

INTERVENTIONS:
Drug: Sterimar Spray — Post-op nasal spray, three times a day
  Other Names: Sterimar nasal seawater spray
  Arms: 1
Drug: Generic homemade nasal saline spray (salt and water) — post op nasal saline spray in syringe, three times a day
  Other Names: generic salt water solution
  Arms: 2

SUMMARY:
Patients undergoing nasal surgery commonly experience a variety of symptoms in the post-operative period including blockage, running, pain, bleeding and reduction in sense of smell. A variety of preparations are currently recommended for symptomatic relief in the post operative period. These include saline irrigations and sniffs, steam inhalations, decongestants and steroid drops.

There is currently no level 1 evidence in literature to support the use of any particular preparation over others in nasal surgical aftercare.

We propose to conduct a single blinded, randomised trial comparing saline sprays vs Sterimar, a commercially available aerosolised isotone saline solution, comparing patients' symptom scores following septal surgery.

The trial will help to establish efficacy and symptom control and advantages of one solution and delivery device over the other.

DETAILED DESCRIPTION:
Project Proposal

Sterimar vs Saline Sprays in nasal surgical aftercare - a blinded, randomised trial.

Gundula Thiel, Andy Evans, Kim Ah-See

Background

Patients undergoing nasal surgery commonly experience a variety of symptoms in the post-operative period including blockage, running, pain, bleeding and reduction in sense of smell. A variety of preparations are currently recommended for symptomatic relief in the post operative period. These include saline irrigations and sniffs, steam inhalations, decongestants and steroid drops. These are intended to reduce swelling and crusting and their resultant symptoms.

There is currently no level 1 evidence in literature to support the use of any particular preparation over others in nasal surgical aftercare.

A recent randomised controlled trial carried out in this department, comparing use of xylometazoline based decongestants vs Sterimar seawater nasal spray, showed a lower pain scoring in the Sterimar group but no other significant differences. This study is as yet unpublished.

Sterimar spray is a spray made from seawater which is diluted to make the solution isotonic.

Traditionally, other forms of Saline sniffs and rinses are also used for the above mentioned applications.

It is easy to make up an isotonic saline solution, using 5 grams of salt (1 teaspoon) for every ½ litre of boiled water. This can then, after cooling off, be applied to the nasal cavities with the help of a standard 10 ml syringe which is provided to the patient at discharge.

As Sterimar is not yet on the hospital formulary, the cost for the treatment is currently borne by the patient. For the duration of the study, patients randomized into the Sterimar group will be provided with the medication free of charge.

We consider it unlikely that patients randomised into the saline spray group will supplement this treatment by buying further saline sprays from the chemist at their own expense.

To establish this and to follow up patients after the trial period, we will establish a research clinic. Patients will be reviewed in a clinic dedicated to patients taking part in this trial approximately 2 weeks after surgery, after completion of the trial period.

The trial will help to establish efficacy and symptom control and advantages of one solution and delivery device over the other.

If home-made saline sprays could be used to similar effect as Sterimar, the cost for this form of surgical aftercare could be lowered significantly, both for the patient and the NHS.

We propose to conduct a single blinded, randomised trial comparing saline sprays vs Sterimar, a commercially available aerosolised isotone saline solution, comparing patients' symptom scores following septal surgery.

The MHRA confirmed that neither the Sterimar nor the home made saline spray are considered Investigational Medicinal Products.

Methodology

Setting

ENT unit, Aberdeen Royal Infirmary, teaching hospital

Inclusions / exclusions

Patients undergoing septoplasty and septoplasty in conjunction with turbinate surgery will be recruited. Those undergoing additional procedures including polypectomy will be excluded, as will all patients whose post-operative recommendations are for steroids or other take home medications that may bias results.

Recruitment

Patients fitting the inclusion criteria will be approached in the Outpatients clinic. The decision for septoplasty +/- turbinate surgery will be made there and consent for the operation will be taken. A patient information sheet will be administered by the lead investigator or other medical staff on the same day, allowing the patient ample time to discuss the matter with relatives and medical staff. Patients will be left to read the information sheet and then re-approached to assess willingness to be included in the trial. The procedure of the trial will be further explained and informed consent to take part will be obtained. Patients will retain the patient information sheet as well as receive a scoring sheet containing visual analogue scales to assess symptoms - pain, running, sense of smell, bleeding, blockage. A questionnaire assessing use of post-operative analgesia for 7 days on a daily basis will also be included.

All these forms will be on appropriately headed paper. A clear explanation of how to complete the assessment sheet will be given. The patient will be approached again on the pre-operative morning and Patients will be randomised using a randomisation schedule generated by NHS Grampian Research & Development Dept.

can withdraw his/her consent to the trial at any time. Randomisation

Patients will be randomised using a randomisation schedule generated by NHS Grampian Research & Development Dept.

Treatment

Based on the randomisation, patients will be given one of either saline sprays or Sterimar Physiological Sea Water Microspray. Instructions regarding use will be given including frequency and technique.

Outcome measures

On the 3rd and 7th postoperative day, patients will complete the symptom assessment sheet judging their symptoms on that day.

The patient should record painkillers needed on the Analgesia Requirement Sheet on a daily basis for 7 days.

The patients will also be provided with an EQ-5D health questionnaire, which is well validated and has referent look up values for populations of ill and healthy patients.

These will be returned in a pre-paid envelope and will be identifiable only by the patients' study number retained in the randomisation program.

Analysis

Visual analogue scales will be analyzed by investigators blinded to which treatment has been administered.

Results will be further analysed comparing scores achieved for those taking saline sniffs and those taking Sterimar. Tests of statistical significance will be performed to establish if either preparation is superior in symptom control. Analgesia use will be taken into consideration.

To select a difference in symptom scores on a visual analogue scale of 10mm or more at the level of significance with 80% power, a sample size of 60 patients is required in each arm of the trial. This is assuming a standard deviation of 19mm, which was demonstrated in the study previously conducted in this department.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing septoplasty and septoplasty in conjuction with turbinate surgery will be recruited.

Exclusion Criteria:

* Those undergoing additional procedures including polypectomy will be excluded, as will all patients whose post-operative recommendations are for steroids or other take home medications that may bias results.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
On the 3rd and 7th postoperative day, patients will judge their symptoms on that day, using VAS. | Day 3 and 7

SECONDARY OUTCOMES:
The patient should record painkillers needed on a daily basis for 7 days and will be provided with an EQ-5D health questionnaire. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kim W Ah-See, MD, FRCS, Principal Investigator — NHS Grampian
Locations (1):
- Department of Otorhinolaryngology, Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom